CLINICAL TRIAL: NCT05001113
Title: Comparison of Safety and Perioperative Outcomes of Subxiphoid Approach Versus Lateral Intercostal Approach Thoracoscopic Thymectomy for Masaoka-Koga I-II Thymoma: A Prospective, Open, Multi-center, Phase II Randomized Controlled Trial
Brief Title: Surgery for Masaoka-Koga I-II Thymoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Zhongshan Hospital (Xiamen), Fudan University (Other); Xuhui Central Hospital, Shanghai (Other); Shanghai Minhang Central Hospital (Other); Shanghai Qingpu Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-454
Record Dates: First submitted 2021-07-12; First posted 2021-08-11 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Thymoma; Masaoka Stage I; Masaoka Stage II
Keywords: thymoma (Masaoka Stage I-II); the subxiphoid approach; the lateral intercostal approach
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the subxiphoid approach thoracoscopic thymectomy (Experimental): The subxiphoid approach thoracoscopic thymectomy is performed in enrolled patients.
  Interventions: Procedure: the subxiphoid approach thoracoscopic thymectomy
- the lateral intercostal approach thoracoscopic thymectomy (Active Comparator): The lateral intercostal approach thoracoscopic thymectomy is performed in enrolled patients.
  Interventions: Procedure: the lateral intercostal approach thoracoscopic thymectomy

INTERVENTIONS:
Procedure: the subxiphoid approach thoracoscopic thymectomy — A 2-cm straight incision was made in the middle of the xiphoid process, the incision was used as a thoracoscope hole, and the xiphoid process could be removed if necessary. The surgeon used the oval forceps to release the left and right soft tissue gaps behind the sternum, from the anterior mediastinum tunnel. Two 0.5 cm extrapleural thoracic ports under the bilateral costal arches were created, and this incision was used as an operation hole. The thread puncture cone with a diameter of 0.5 cm was placed under the guidance of the finger.
  Other Names: SATT
  Arms: the subxiphoid approach thoracoscopic thymectomy
Procedure: the lateral intercostal approach thoracoscopic thymectomy — Right-side approach: Use the left supine position. The observing port was created at the right axillary midline line in the fourth intercostal space, and the other two ports were made as to the operation hole along the anterior axillary lines in the third and fifth intercostal spaces.
  Left-side approach: Use the right supine position. The observing port was created at the left axillary midline line in the fourth intercostal space, and the other two ports were made as to the operation hole along the anterior axillary lines in the third and fifth intercostal spaces.
  Other Names: LATT
  Arms: the lateral intercostal approach thoracoscopic thymectomy

SUMMARY:
The purpose of this study was to evaluate the safety and perioperative outcomes of the subxiphoid approach versus the lateral intercostal approach thoracoscopic thymectomy for Masaoka-Koga I-II thymoma.

DETAILED DESCRIPTION:
It is a multi-center, open, prospective randomized phase II&III clinical trial sponsored by Shanghai Zhongshan Hospital with other four hospitals in China participating in. 100 patients with thymoma (Masaoka-Koga I-II ) diagnosed by enhanced computed tomography were recruited and randomly assigned into the subxiphoid approach thoracoscopic thymectomy (SATT group) and the lateral intercostal approach thoracoscopic thymectomy (LATT group) according to the proportion of 1:1. The safety and perioperative outcomes are compared between the two surgical regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Thymoma was diagnosed by chest enhanced CT (clinical stage: Masaoka Koga I-II);
2. The patients whose tumor diameter was <6 cm;
3. The patients with age ≥ 18 and ≤ 75 years old, the estimated survival time should be over 12 months;
4. ASA grade：1-2;
5. The patients should have no functional disorders in main organs.;
6. The patients should be able to understand our research and sign the informed consent.

Exclusion Criteria:

1. Imaging examination showed that the tumor had invasion of surrounding organs, pleural or pericardial dissemination, lymphatic or hematogenous metastasis;
2. Patients with myasthenia gravis;
3. Patients had undergone a sternotomy;
4. The patients have proved history of congestive heart failure, angina without good control with medicine; ECG-proved penetrating myocardial infarction; hypertension with bad control; valvulopathy with clinical significance; arrhythmia with high risk and out of control;
5. The patients have severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under treatment of thrombolysis or anticoagulant therapy;
6. Female who is positive for serum pregnancy test or during lactation period;
7. The patients have history of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation;
8. The patients have history of peripheral nerve system disorders, obvious mental disorders or central nerve system disorders;
9. The patients attend other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Dosage of analgesic medication after surgery | Up to the date of hospital discharge since the data of completion of surgery, up to 7 days
  The dosage of postoperative analgesic medication was the sum of the dosage of analgesics used for managing the pain of the patient after surgery. The analgesic medication includes analgesics in patient-controlled epidural analgesia (PCIA), injections, and oral medication.
Visual Analog Scales scores for postoperative pain | Up to the date of hospital discharge since the data of completion of surgery, up to 7 days
  The postoperative pain was evaluated for every enrolled patient by using the Visual Analog Scales (VAS).
  VAS: it typically asks a patient to place a mark on a line indicating the level of pain from 0 to 10. Zero indicates the absence of pain, while 10 represents the most intense pain possible.
Postoperative hospital stay | Up to the date of meeting the criteria of hospital discharge since the data of surgery, up to 1 month
  Postoperative hospital stay is the duration for every enrolled patient until the date of meeting the criteria of hospital discharge since the date of surgery.
  The criteria of hospital discharge were defined as with the volume of postoperative drainage < 200 ml/day, a normal chest X-ray, and good physical condition.

SECONDARY OUTCOMES:
Operative time | The duration until the finish of surgery since the start of the surgery, up to 5 hours
  Operative time was defined as the time between the start of the surgery (incision) and the finish of surgery (closure of the skin).
Perioperative blood loss | The duration until the finish of surgery since the start of the surgery, up to 5 hours
  The volume of bleeding during the surgery.
Rate of conversion to open thoracotomy | Up to the end of follow-up since the date of randomization, up to 6 months.
  It was the proportion of operations with unplanned conversion to thoracotomy in total operations in every group. The formula： Number (operations with unplanned conversion to thoracotomy in every group) / 50 * 100%.
Volume of postoperative drainage | Up to the date of removal of drainage equipment since the data of completion of surgery, up to 7 days
  The volume of postoperative drainage of the patient was the sum of his daily drainage volume after the surgery. The types of drainage equipment include the thorax close drainage equipment and the unidirectional negative-pressure drainage ball.
Postoperative treatment-related complications | Up to the date of hospital discharge since the data of completion of surgery, up to 7 days.
  Number and severity of adverse events that are related to the treatment of each patient. Postoperative treatment-related complications were assessed by the Clavien-Dindo Classification. Treatment-related adverse events as assessed by CTCAE v5.0.
Chronic postsurgical pain | Up to the end of follow-up since the date of hospital discharge, up to 6 months.
  An updated definition of chronic postsurgical pain (CPSP) was proposed by Werner and Kongsgaard in 2014.
  The proposed definition of CPSP was "pain persisting at least three months after surgery, that was not present before surgery, or that had different characteristics or increased intensity from preoperative pain, localized to the surgical site or a referred area, and other possible causes of the pain were excluded (e.g., cancer recurrence, infection)".
EORTC QLQ-C30 score for overall quality of life | Up to the end of follow-up since the date of randomization, up to 6 months.
  Overall quality of life is respectively evaluated at randomization and 1 month, 3 month, 6 month after surgery among patients by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 Scale (EORTC QLQ-C30) (V3.0).
  The minimum value of EORTC QLQ-C30 score was 0，and the maximum was 100. Zero indicates the worst quality of life, while 100 represents the best quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
According to the regulations on the management of human genetic resources of the People's Republic of China, we will not be able to share Individual Participant Data